CLINICAL TRIAL: NCT04364009
Title: Efficacy and Safety of ANAkinra During Adult " COVID-19 " With Aggravating Respiratory Symptoms: a Multicenter Open-label Controlled Randomized Trial
Brief Title: Anakinra for COVID-19 Respiratory Symptoms
Acronym: ANACONDA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Efficiency and safety reasons
Sponsor: University Hospital, Tours (Other)
Collaborators: INSERM CIC-P 1415, University Hospital Center of Tours (Unknown); Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANACONDA-COVID-19; 2020-001734-36 (EudraCT Number); DR200111 (Other: University Hospital of Tours)
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Infection; ANAKINRA Treatment; Optimized Standard of Care (oSOC)
MeSH Terms: conditions — COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: ANACONDA study is a French multicentre, open-label, randomized, controlled superiority trial comparing the administration of optimized standard of care and Anakinra versus optimized standard of care alone in patients hospitalized in a medical unit with COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized Standard of Care (oSOC) (Active Comparator): The control group will receive optimized standard of care alone, including all treatments authorized for COVID-19 by the French Health Ministry and/or the center COVID-19 therapeutic committees at inclusion and during the follow-up.
  Interventions: Drug: oSOC
- Anakinra plus Optimized Standard of Care (oSOC) (Experimental): The experimental group will receive Anakinra plus optimized Standard of Care. The patients will receive Intravenous injection (IV) of Anakinra 400mg/day (100mg IV every 6 hours) at Day 1, 2 and 3. From Day 4 to Day 10, the patient will receive IV injection of Anakinra 200mg/day (100mg every 12 hours). The total duration of Anakinra is 10 Days
  Interventions: Drug: Anakinra plus oSOC

INTERVENTIONS:
Drug: Anakinra plus oSOC — Anakinra plus Optimized Standard of Care (oSOC) on the condition of patients with COVID-19 infection and worsening respiratory symptoms.
  The patients will receive intraveinous injection of Anakinra 400mg from Day 1 to Day 3 (two injections of 100 mg each 12 hours) and 200mg the remaining 7 days. The total duration of Anakinra is 10 Days. Efficient dosage of Anakinra as previously described will be continued until Day 10
  Arms: Anakinra plus Optimized Standard of Care (oSOC)
Drug: oSOC — Optimized Standard of Care (oSOC) on the condition of patients with COVID-19 infection and worsening respiratory symptoms.
  Arms: Optimized Standard of Care (oSOC)

SUMMARY:
The main objective of the ANACONDA-COVID-19 trial is to assess the efficacy of Anakinra + optimized Standard of Care (oSOC) as compared to oSOC alone on the condition of patients with COVID-19 infection and worsening respiratory symptoms. Success defined as patient alive and free of invasive mechanical ventilation (IMV) and free of Extracorporeal Membrane Oxygenation (ECMO) at Day 14.

ELIGIBILITY:
Inclusion criteria:

* Male or female≥ 18 years of age
* Written informed consent of the patient or a proxy
* Ability for participant to comply with the requirements of the study
* Hospitalized patient with COVID-19 defined as

  * Positive SARS-CoV2 RT-PCR
  * Or typical COVID-19 Radiographic infiltrates on the CT scan (peripheral ground glass without lung cavitation, lymphadenopathy, or pulmonary nodules) other non COVID-19 diagnosis ruled out.
* Patient with respiratory symptoms and requirement of oxygen therapy as defined:

  * Oxygen therapy >= 4L/min to maintain Sp02>92% and respiratory rate >=24/min.
  * Or patients under oxygen >= 1L/min and presenting worsening of oxygen requirement defined by an increase of oxygen therapy >= 2L/min to maintain Sp02>92%.
* Inflammatory component C-Reactive Protein ≥ 50mg/L.
* Patients within the first 20 days from the onset of the first COVID-19 symptoms
* Probabilistic antibiotics therapy according to local practice

Non-inclusion criteria:

* Respiratory failure related to other cause than COVID-19
* Patients requiring mechanical ventilation at inclusion or requiring oxygen therapy equal or more than 11 liters per min to maintain Sp02>92%
* Infectious diseases such as severe bacterial infections, aspergillosis, HIV, active HCV, active HBV, active tuberculosis
* Contra indication to anti-IL1 receptor

  * Known hypersensitivity to Anakinra
  * Absolute neutrophil count (ANC)< 1500/mm3
  * Liver cirrhosis Child-Pugh Score C
  * Live or attenuated vaccine in the past 8 weeks
  * Pregnant or breast-feeding women
* Patients with either legally protected status or who have been deprived of their freedom
* Patient included in other interventional therapeutic research (e.g. = concurrent participation in French CoVID-19 is accepted)
* Patients who have received previous treatment by anti-IL6R, anti-IL-6, anti-IL1R, anti-IL1 or anti-TNFα within 21 days preceding inclusion
* Absence of Health Insurance
* Existence of any life-threatening co-morbidity or any other medical condition which,in the opinion of the investigator, makes the patient unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Treatment success | After 14 days of treatment
  The primary endpoint is treatment success at Day 14, defined as a patient alive and not requiring any of the following: Invasive mechanical ventilation (IMV) or Extracorporeal membrane oxygenation (ECMO).

SECONDARY OUTCOMES:
Treatment success | After 3 days, 10 days and 28 days of treatment
  Defined as a patient alive and not requiring any of the following: Invasive mechanical ventilation (IMV) or Extracorporeal membrane oxygenation (ECMO).
OMS progression scale (on a 7 point ordinal scale) | After 3 days, 10 days, 14 days and 28 days of treatment
  1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities; 3. Hospitalized, not requiring supplemental oxygen; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;6. Hospitalized, on invasive mechanical ventilation or ECMO;7. Death.
Overall survival | After 3 days, 10 days, 14 days and 28 days of treatment
  Overall survival
Time to ICU admission | Up to 28 days
  Time to ICU admission
Time to ventilatory support | Up to 28 days
  Time to ventilatory support : extracorporeal membrane oxygenation (ECMO), invasive mechanical ventilation, non-invasive ventilation, high flow oxygen therapy)
Change in National Early Warning Score (NEW)from baseline to Day 3, Day 10, Day 14 and Day 28 | After 3 days, 10 days, 14 days and 28 days of treatment
  The National Early Warning Score (NEWS) determines the degree of illness of a patient using six physiological findings and one observation. Score from 0 to 20, 0 mean a worse outcome, 20 mean a better outcome
Change in inflammatory parameter | From baseline to Day 3, Day 10, Day 14 and Day 28
  C-reactive proteine (mg/L)
Change in inflammatory parameter | From baseline to Day 3, Day 10, Day 14 and Day 28
  ferritin (ng/mL)
Change in inflammatory parameter | From baseline to Day 3, Day 10, Day 14 and Day 28
  lymphocyte count (G/L)
Change in inflammatory parameter | From baseline to Day 3, Day 10, Day 14 and Day 28
  fibrinogen (g/l)
Hospital length of stay | Up to 28 days
  Hospital length of stay
ICU parameter | Up to 28 days
  Need for Vasopressors (yes or no)
ICU parameter | Up to 28 days
  Evolution of SpO2/FIO2 ratio (no unit)
ICU parameter | Up to 28 days
  Evolution of PaO2/FiO2 ratio (no unit)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 28 days
  Occurrence of serious adverse events during the study, including infection (bacterial, parasitic, mycotic and viral infection), septic shock, Ankanira hypersensitivity, hepatic damages (SGOT/SGPT, alkaline phosphatase, gammaGT) and neutropenia (Blood count).
Predictors of efficacy of Anakinra | After 14 days of treatment
  The correlation between several of clinical parameters at inclusion (including level of oxygen requirement (saturation), respiratory rate (per min), temperature (°C)…), biological parameters :including, CRP (mg/L), ferritin (µg/L), LDH (UI/L), lymphocyte count (G/L), eosinophil count (G/L), Ddimers (ng/mM), platelet count (G/L), polymorphonuclear count (G/L)...with the primary end point will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra AUDEMARD-VERGER, MD-PhD, Study Director — University Hospital of Tours
Locations (1):
- CHRU de TOURS, Tours, France

IPD SHARING:
Plan to Share IPD: No